CLINICAL TRIAL: NCT06506123
Title: Automated Detection and Classification of Patient-Ventilator Dyssynchrony With a Machine Learning Algorithm
Brief Title: Patient-Ventilator Dyssynchrony Detection With a Machine Learning Algorithm
Status: Recruiting | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Magnamed Tecnologia Medica S/A (Unknown)
Responsible Party: Sponsor
Other Study IDs: CAAE 78855824.7.0000.0068
Record Dates: First submitted 2024-05-24; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Failure
Keywords: mechanical ventilation; artificial intelligence
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Artificial Intelligence Detection and Classification of Patient-Ventilator Dyssynchronies: This is a single arm study, since all subjects included will be exposed to both diagnostic methods (artificial intelligence and experts). The proposed diagnostic method is a machine learning algorithm integrated in the mechanical ventilator FlexiMag Max 700 (Magnamed, Brazil), which will continuously record data from mechanical ventilation of included subjects for a time period of up to 72 hours. The gold-standard involves esophageal pressure waveform recording and offline analysis by experts.
  Interventions: Device: Artificial Intelligence Detection and Classification of Patient-Ventilator Dyssynchronies

INTERVENTIONS:
Device: Artificial Intelligence Detection and Classification of Patient-Ventilator Dyssynchronies — Machine learning algorithm to detect and classify patient-ventilator dyssynchronies, which is integrated in the mechanical ventilator (Fleximag Max, Magnamed, Brazil).

SUMMARY:
This is a diagnostic study aiming to compare accuracy to detect and classify patient-ventilator dyssynchronies by a machine learning algorithm, compared to the gold-standard defined as dyssynchronies diagnosed and classified by mechanical ventilator and esophageal pressure waveforms analyzed by experts.

The main question of this study is:

• Are patient-ventilator dyssynchronies accurately detected and classified by an artificial intelligence algorithm when compared to experts analyzing esophageal pressure and mechanical ventilator waveforms?

DETAILED DESCRIPTION:
This is a diagnostic, observational study, aiming to assess patient-ventilator dyssynchrony automated detection and classification by a machine learning algorithm. Accuracy of the machine learning algorithm will be compared with the gold-standard, defined as dyssynchronies detected and classified by mechanical ventilation experts.

Experts will analyzed airway pressure, flow, volume and esophageal pressure waveforms to detect and classify dyssynchronies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects under assisted or assist-controlled mechanical ventilation and monitored with esophageal pressure balloon.

Exclusion Criteria:

* Refusal from patient's family or attending physician

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult subjects under mechanical ventilation, with an assisted or assist-controlled mode, who are monitored with an esophageal pressure balloon due to clinical indication are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-05-25 (Actual); Primary Completion 2025-05-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of the Artificial Intelligence algorithm | 3 days
  Sensitivity, specificity, positive predictive value, negative predictive value of the artificial intelligence algorithm to detect and classify patient-ventilator dyssynchronies. These accuracy indexes will be estimated for each kind of dyssinchrony: ineffective effort, autotriggering, double triggering, reverse triggering, reverse triggering with a double cycle

SECONDARY OUTCOMES:
Pendelluft detection | 3 days
  Percentage of cycles with pendelluft detected with the artificial intelligence algorithm compared to the percentage of cycles with pendelluft detected with the esophageal pressure

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo LV Costa, MD, PhD, Study Director — University of Sao Paulo
Locations (1):
- Heart Institute, University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amato MB, Barbas CS, Medeiros DM, Magaldi RB, Schettino GP, Lorenzi-Filho G, Kairalla RA, Deheinzelin D, Munoz C, Oliveira R, Takagaki TY, Carvalho CR. Effect of a protective-ventilation strategy on mortality in the acute respiratory distress syndrome. N Engl J Med. 1998 Feb 5;338(6):347-54. doi: 10.1056/NEJM199802053380602. PMID 9449727
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Sousa MLEA, Magrans R, Hayashi FK, Blanch L, Kacmarek RM, Ferreira JC. Clusters of Double Triggering Impact Clinical Outcomes: Insights From the EPIdemiology of Patient-Ventilator aSYNChrony (EPISYNC) Cohort Study. Crit Care Med. 2021 Sep 1;49(9):1460-1469. doi: 10.1097/CCM.0000000000005029. PMID 33883458
- [Background] Sousa MLA, Magrans R, Hayashi FK, Blanch L, Kacmarek RM, Ferreira JC. Predictors of asynchronies during assisted ventilation and its impact on clinical outcomes: The EPISYNC cohort study. J Crit Care. 2020 Jun;57:30-35. doi: 10.1016/j.jcrc.2020.01.023. Epub 2020 Jan 21. PMID 32032901
- [Background] Blanch L, Villagra A, Sales B, Montanya J, Lucangelo U, Lujan M, Garcia-Esquirol O, Chacon E, Estruga A, Oliva JC, Hernandez-Abadia A, Albaiceta GM, Fernandez-Mondejar E, Fernandez R, Lopez-Aguilar J, Villar J, Murias G, Kacmarek RM. Asynchronies during mechanical ventilation are associated with mortality. Intensive Care Med. 2015 Apr;41(4):633-41. doi: 10.1007/s00134-015-3692-6. Epub 2015 Feb 19. PMID 25693449
- [Background] LeCun Y, Bengio Y, Hinton G. Deep learning. Nature. 2015 May 28;521(7553):436-44. doi: 10.1038/nature14539. PMID 26017442